CLINICAL TRIAL: NCT02253771
Title: Shockwave Therapy for Acute Low Back Pain: a Randomized Placebo-controlled Clinical Trial
Brief Title: Shockwave Therapy for Acute Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Responsible Party: Principal Investigator, Niklas Deventer, Dr. med. Niklas Deventer, University Hospital Muenster
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Orth-001
Record Dates: First submitted 2014-08-31; First posted 2014-10-01 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Acute Low Back Pain (Low Back Pain for Less Than 3 Months)
MeSH Terms: interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- shockwave therapy (Experimental): shockwave therapy
  Interventions: Device: shockwave therapy
- Placebo treatment (Placebo Comparator): sham shockwave therapy by an identically looking device without any function
  Interventions: Device: placebo shockwave therapy

INTERVENTIONS:
Device: shockwave therapy — Shockwave therapy with 2000 impulses/treatment at 12 Hz; 8 treatment over 4 weeks, twice a week
  Other Names: EMS Swiss Dolorclast® Classic (EMS Electro Medical Systems S.a.); CE Certificate: 0124
  Arms: shockwave therapy
Device: placebo shockwave therapy — sham shockwave therapy by an identically looking device without any function
  Arms: Placebo treatment

SUMMARY:
The purpose of this study is to determine whether shockwave therapy is more effective in the treatment of unspecific acute low back pain than sham therapy.

60 patients with acute low back pain will be recruited to a single-blinded, randomized, placebo-controlled trial. They are randomized to receive either shockwave therapy or sham treatment by a identically looking device for 4 weeks, twice a week. Additionally patients receive physiotherapy twice a week and are allowed to take an anti-inflammatory drug, if necessary for even 4 weeks. The primary outcome variable will be measured at day 0, every week during treatment (day 7; 14; 21 and 28) and up to 4 weeks after the last treatment. The clinical outcome will be primarily measured by pain intensity using a visual analogue scale. Secondary outcome measures are Oswestry Disability Index, Beck's Pain Depression Scale, Roland Morris Disability Questionnaire and the EQ-5D. Data will be analysed for the difference in change of scores between groups using one-way t-test.

ELIGIBILITY:
Inclusion Criteria:

low back pain for less than 3 months

Exclusion Criteria:

* Patients with relevant leg pain
* Patients with spine operations in the past
* neurologic symptoms
* scoliosis with Cobb angle > 10°
* Patients experienced in shock wave therapy
* Patientes with ongoing therapy with blood diluting drugs such as phenprocumon
* Patients with osteoporosis
* Patients with back pain after trauma
* Patients with infective diseases or tumor diseases
* Patients with relevant psychological diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2018-09-13 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Change in pain, using visual analogue scale (VAS) | Day 0; 7; 14; 21; 28, after 6 and 8 weeks.
  Change in pain, using visual analogue scale (VAS 1-10)

SECONDARY OUTCOMES:
Change in other clinical questionnaires (Oswestry disability Index) | day 0; 7; 14; 21, after 6 and 8 weeks.
  Oswestry disability Index
Change in other clinical questionnaires (Beck's depression scale) | day 0; 7; 14; 21, after 6 and 8 weeks.
  Beck's depression scale
Change in other clinical questionnaires (EQ-5D) | day 0; 7; 14; 21, after 6 and 8 weeks.
  EQ-5D
Change in other clinical questionnaires (Roland-Morris-Score) | day 0; 7; 14; 21, after 6 and 8 weeks.
  Roland-Morris-Score

CONTACTS AND LOCATIONS:
Overall Officials: Niklas Deventer, Dr. med., Principal Investigator — Universitätsklinikum Münster, Klinik für Allgemeine Orthopädie und Tumororthopädie; Tobias Schulte, Prof. Dr. med., Study Director — Department of Orthopaedics and Trauma Surgery, University Hospital, Ruhr University Bochum; Tobias Lange, Dr. med., MBA, Principal Investigator — Department of Orthopaedics and Trauma Surgery, University Hospital, Ruhr University Bochum
Locations (1):
- Universitätsklinikum Münster, Klinik für Allgemeine Orthopädie und Tumororthopädie, Münster, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Barker KL, Elliott CJ, Sackley CM, Fairbank JC. Treatment of chronic back pain by sensory discrimination training. A Phase I RCT of a novel device (FairMed) vs. TENS. BMC Musculoskelet Disord. 2008 Jun 28;9:97. doi: 10.1186/1471-2474-9-97. PMID 18588702
- [Background] Seco J, Kovacs FM, Urrutia G. The efficacy, safety, effectiveness, and cost-effectiveness of ultrasound and shock wave therapies for low back pain: a systematic review. Spine J. 2011 Oct;11(10):966-77. doi: 10.1016/j.spinee.2011.02.002. Epub 2011 Apr 9. PMID 21482199